CLINICAL TRIAL: NCT03994250
Title: Kinematic Alignment Compared to Mechanical Alignment Techniques for Total Knee Replacement Surgery (KARMA)
Acronym: KARMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Robert Jones and Agnes Hunt Orthopaedic and District NHS Trust (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: RL1 643
Record Dates: First submitted 2019-01-15; First posted 2019-06-21 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2020-03

CONDITIONS: Osteo Arthritis Knee
Keywords: kinematic; mechanical; total knee replacement

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kinematic Arm (Active Comparator): Kinematic Alignment for TKR surgery
  Interventions: Other: Kinematic Alignment for total knee replacement surgery
- Control Arm (Placebo Comparator): Mechanical alignment for TKR surgery
  Interventions: Other: Mechanical Alignment for total knee replacement surgery

INTERVENTIONS:
Other: Kinematic Alignment for total knee replacement surgery — Using Kinematic Alignment for total knee replacement surgery
  Other Names: Kinematic Arm
  Arms: Kinematic Arm
Other: Mechanical Alignment for total knee replacement surgery — Using mechanical alignment for total knee replacement surgery
  Other Names: Control Arm
  Arms: Control Arm

SUMMARY:
Total knee replacement (TKR) is a bony and soft-tissue procedure and much attention has been given to the alignment of the components, which is relatively easy to quantify. Recently, substantial healthcare resources have been devoted to the development and use of computer navigation and patient-specific instrumentation systems that achieve neutral mechanical alignment. However the conventional assumption that mechanically aligned TKR leads to the best implant survival has been brought into doubt. Although mechanically aligned TKR improves function, 20 % of patients remain dissatisfied according to reports from Canada, England and Wales.

In an attempt to improve patient satisfaction recent developments have included the individualization of component alignment with the goal of achieving pre-arthritic alignment through restoration of the axes of rotation, a technique called kinematic alignment (KA). The outcomes of kinematic alignment have been assessed in case series but so far only one randomised controlled trial (RCT) [Digital Object Identifier (DOI)10.1302/0301-620X.96B7.32812 Published 1 July 2014] undertaken in the USA has compared the clinical results of kinematic alignment using patient-specific instruments with the traditional technique of mechanical alignment, demonstrating a substantial benefit in postoperative patient pain relief and function. Therefore, for direct comparison between kinematic aligned and mechanically aligned surgical techniques for total knee replacement, the investigators would like to undertake a pilot study prior to a larger RCT and recruit a cohort of 15 patients undergoing kinematical aligned TKR. The investigators will use the same device as was used in a previous mechanically aligned study undertaken at our hospital (REC ref: 12/NE/0293 Attune, DePuy, Warsaw IN, in 35 patients based on the same eligibility criteria who will act as controls), which will allow the opportunity to estimate the standard deviation in the control arm in preparation for the larger RCT.

DETAILED DESCRIPTION:
In order to be able to undertake a randomized controlled trial (RCT) comparing the efficacy of kinematic alignment versus conventional mechanical alignment for total knee replacement a robust assessment of the expected standard deviation of the primary outcome measure (Oxford Knee Score [OKS]) in both arms of the proposed RCT must be undertaken, hence this pilot study.

To determine whether there are improved postoperative outcomes in the investigative arm using the following patient reported outcomes: Knee Implant Performance (PKIP - pre and post surgical), Knee Injury and Osteoarthritis Outcome Score (KOOS), Knee Society Score (KSS), Knee Noise and Front of Knee Pain Score and Quality of Life score EQ-5D which will be completed at baseline(pre-operatively) and post-operatively at 6 weeks (normal clinical follow up), 1 year (normal clinical follow up) and 2 years. In addition, x-rays of the knee (AP, lateral & skyline) will be taken at the same time. These outcomes are identical to the data collected in the previous mechanically aligned study which will be used as the control arm.

Much attention has been given to the alignment of the components in total knee replacement (TKR) and this is relatively easy to quantify, particularly in the coronal plane. However, due to the development and use of computer navigation and patient-specific instrumentation systems that achieve neutral mechanical alignment, the conventional assumption that mechanically aligned TKR leads to the best implant survival has been brought into doubt. Although mechanically aligned TKR improves function, 20 % of patients remain dissatisfied according to reports from Canada, England and Wales. The relationship between in-range and varus (turned inward toward the mid line of the body to an abnormal degree) and valgus (turned outward) outlier categories of the limb and implant survival of a primary total knee replacement is weak at 15 years. Leaving a limb, knee, or tibial component within a natural range of varus does not reduce implant survival at 3, 5, 7, and 10 years.

With the development of individualization of component alignment and the goal of achieving pre-arthritic alignment through restoration of the axes of rotation, the kinematic alignment technique has shown in case series and one RCT in the USA a substantial benefit in postoperative patient pain relief and function.

For direct comparison between kinematic aligned and mechanically aligned surgical techniques for total knee replacement, the investigators will conduct a pilot study prior to a larger RCT and recruit a cohort of 15 patients undergoing kinematic aligned TKR. The investigators will use the same device as was used in a previous mechanically aligned study undertaken at our hospital (REC ref: 12/NE/0293 Attune, DePuy, Warsaw IN, in 35 patients based on the same eligibility criteria who will act as controls), which will allow the opportunity to estimate the standard deviation in the control arm in preparation for the larger RCT.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between the age of 22 and 80 years inclusive
* Diagnosis of non-inflammatory degenerative joint disease
* Suitable candidate for cemented primary total knee arthroplasty
* Voluntary, informed consent to participate in the study
* Subject is not currently bedridden
* Able to understand (in the opinion of the clinical investigator) the clinical investigation and co-operate with clinical investigations
* Subject is able to comfortably speak, read and understand questions

Exclusion Criteria:

* Females who are pregnant or lactating
* Contralateral knee already enrolled in the study
* Previous partial knee replacement (unicompartmental, bicompartmental or patellofemoral joint replacement), patellectomy, high tibial osteotomy or primary TKA in affected knee
* Contralateral amputation
* Currently experiencing radicular pain from the spine
* Participated in a study with an investigational product in the last 3 months
* Currently involved in any personal injury litigation, medical-legal or workers compensation claims
* Known drug or alcohol abuser or a psychological disorder that could affect their ability to complete patient reported questionnaires
* Diagnosed with fibromyalgia that is currently being treated with prescription medication
* Significant neurological or musculoskeletal disorders or disease that may adversely affect gait or weight bearing (e.g. muscular dystrophy, multiple sclerosis, Charcot disease)
* Suffering with inflammatory arthritis (e.g. rheumatoid arthritis, juvenile rheumatoid arthritis,psoriatic arthritis, systemic lupus erythematosus
* Medical condition with less than 2 years life expectancy

Ages: 22 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-02-10 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Oxford Knee Score measuring current mobility and knee pain | Up to 2 weeks prior to surgery
  Questionnaire, highest score 48 indicates good mobility and no knee pain
Oxford Knee Score | up to 6 weeks post surgery
  Questionnaire, highest score 48 indicates good mobility and no knee pain
Oxford Knee Score | up to 1 year post surgery
  Questionnaire, highest score 48 indicates good mobility and no knee pain
Oxford Knee Score | up to 2 years post surgery
  Questionnaire, highest score 48 indicates good mobility and no knee pain

SECONDARY OUTCOMES:
Knee Injury and Osteoarthritis Outcome Score (KOOS) | Up to 2 weeks prior to surgery
  Questionnaire, highest score 100% to assess the patient's opinion about their knee and associated problems
Knee Injury and Osteoarthritis Outcome Score (KOOS) | up to 6 weeks post surgery
  Questionnaire, highest score 100% to assess the patient's opinion about their knee and associated problems
Knee Injury and Osteoarthritis Outcome Score (KOOS) | up to 1 year post surgery
  Questionnaire, highest score 100% to assess the patient's opinion about their knee and associated problems
Knee Injury and Osteoarthritis Outcome Score (KOOS) | up to 2 years post surgery
  Questionnaire, highest score 100% to assess the patient's opinion about their knee and associated problems
Knee Society Score (KSS) | Up to 2 weeks Prior to surgery
  Questionnaire, +80 Excellent, -60 Poor, Alignment, stability, joint motion of knee, symptoms, patient satisfaction, patient expectations, functional activities, normal, advanced and discretionary activities
Knee Society Score (KSS) | Up to 6 weeks post surgery
  Questionnaire, +80 Excellent, -60 Poor, Alignment, stability, joint motion of knee, symptoms, patient satisfaction, patient expectations, functional activities, normal, advanced and discretionary activities
Knee Society Score (KSS) | Up to 1 year post surgery
  Questionnaire, +80 Excellent, -60 Poor, Alignment, stability, joint motion of knee, symptoms, patient satisfaction, patient expectations, functional activities, normal, advanced and discretionary activities
Knee Society Score (KSS) | Up to 2 years post surgery
  Questionnaire, +80 Excellent, -60 Poor, Alignment, stability, joint motion of knee, symptoms, patient satisfaction, patient expectations, functional activities, normal, advanced and discretionary activities
Quality of Life Score (EQ-5D) | Up to 2 weeks Prior to surgery
  Questionnaire, 1.000 excellent, -0.5 poor, patient mobility, self-care, usual activities, pain/discomfort, anxiety/Depression and patient's view of their health.
Quality of Life Score (EQ-5D) | Up to 6 weeks post surgery
  Questionnaire, 1.000 excellent, -0.5 poor, patient mobility, self-care, usual activities, pain/discomfort, anxiety/Depression and patient's view of their health.
Quality of Life Score (EQ-5D) | Up to 1 year post surgery
  Questionnaire, 1.000 excellent, -0.5 poor, patient mobility, self-care, usual activities, pain/discomfort, anxiety/Depression and patient's view of their health.
Quality of Life Score (EQ-5D) | Up to 2 years post surgery
  Questionnaire, 1.000 excellent, -0.5 poor, patient mobility, self-care, usual activities, pain/discomfort, anxiety/Depression and patient's view of their health.
Knee Noise and Front of Knee Pain | Up to 2 weeks prior to surgery
  Questionnaire detecting crepitus in the knees which may be caused by a meniscus tear or chondromalacia patellais, for example, a dull ache behind the kneecap
Knee Noise and Front of Knee Pain | Up to 6 weeks post surgery
  Questionnaire detecting crepitus in the knees which may be caused by a meniscus tear or chondromalacia patellais, for example, a dull ache behind the kneecap
Knee Noise and Front of Knee Pain | Up to 1 year post surgery
  Questionnaire detecting crepitus in the knees which may be caused by a meniscus tear or chondromalacia patellais, for example, a dull ache behind the kneecap
Knee Noise and Front of Knee Pain | Up to 2 years post surgery
  Questionnaire detecting crepitus in the knees which may be caused by a meniscus tear or chondromalacia patellais, for example, a dull ache behind the kneecap
Patient Knee Implant Performance | Up to 2 weeks Prior to surgery
  Questionnaire, 0 - 100 (higher better knee function) 4 subscales (Confidence, stability, modify activities and satisfaction) each with score of 0 - 10 (latter better knee function)
Patient Knee Implant Performance | Up to 6 weeks post surgery
  Questionnaire, 0 - 100 (higher better knee function) 4 subscales (Confidence, stability, modify activities and satisfaction) each with score of 0 - 10 (latter better knee function)
Patient Knee Implant Performance | Up to 1 year post surgery
  Questionnaire, 0 - 100 (higher better knee function) 4 subscales (Confidence, stability, modify activities and satisfaction) each with score of 0 - 10 (latter better knee function)
Patient Knee Implant Performance | Up to 2 years post surgery
  Questionnaire, 0 - 100 (higher better knee function) 4 subscales (Confidence, stability, modify activities and satisfaction) each with score of 0 - 10 (latter better knee function)

CONTACTS AND LOCATIONS:
Overall Officials: JP Whittaker, FRCS, Principal Investigator — Consultant Orthopaedic Surgeon
Locations (1):
- Robert Jones & Agnes Hunt Orthopaedic Hospital NHS Trust, Gobowen, Shropshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No